CLINICAL TRIAL: NCT00555360
Title: Enhancing Caregiver Support for Patients With Heart Failure
Brief Title: Enhancing Caregiver Support for Heart Failure Patients: the CarePartner Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IIR 07-185
Record Dates: First submitted 2007-11-06; First posted 2007-11-08 (Estimated); Results first posted 2015-09-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-08

CONDITIONS: Heart Failure, Congestive
Keywords: Health Information Technology; Patient Care Management; Self Care; Quality of Life; Family or non-Family Informal Caregivers
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Veterans with heart failure that can identify an out-of-home informal caregiver
  Interventions: Behavioral: HITCM+CP
- Arm 2 (Active Comparator): Veterans with heart failure that can identify an out-of-home informal caregiver
  Interventions: Behavioral: HITCM only

INTERVENTIONS:
Behavioral: HITCM+CP — Weekly automated assessment calls with follow-up by a care manager and a CarePartner for 12 months. Baseline, 6-month and 12-month follow-up.
  Arms: Arm 1
Behavioral: HITCM only — Weekly automated assessment calls with follow-up by a care manager for 12 months. Baseline, 6-month and 12-month follow-up.
  Arms: Arm 2

SUMMARY:
Informal caregivers, assisted by health information technology may help to fill the gaps in VA care management of heart failure patients by enhancing support for patients' treatment adherence, behavior changes, and symptom monitoring.

DETAILED DESCRIPTION:
Background: Heart failure (HF) is a leading cause of preventable hospitalization and death in the VA and many patients fall short of self-care goals. Numerous efficacy trials have shown that HF care management supported by health information technology (i.e., HITCM) can improve patients' outcomes, although VA care managers in 'real-world' health systems are often overwhelmed by the need to provide monitoring and behavior change services. Informal caregivers may help to fill the gaps in VA care management and enhance support for patients' treatment adherence, behavior changes, and symptom monitoring. The challenge will be to identify ways to leverage assistance from informal caregivers (ICGs) who lack the resources to fill this role effectively.

Objectives: We will evaluate the impact of extending the reach of HITCM by incorporating a protocol-driven model for improved monitoring and self-management support by a CarePartner (CP). CPs will be adult children or friends living outside the patient's home who are willing to play a structured role to support self-care. The specific aims of the trial are: (1) to determine whether an intervention that uses automated patient monitoring and behavior change calls with follow-up to HF patients' care manager and CP (HITCM+CP) improves key patient-centered outcomes relative to a system that only uses the same technology to support patients' care management (HITCM-only). Outcomes of interest include patients' health-related quality of life, mental health, health service use, and mortality risk; (2) to evaluate the impact of HITCM+CP on patients' self-care behaviors compared to HITCM-only; and (3) to determine whether the intervention increases the quality and quantity of support for HF patients' self-care compared to HITCM-only.

Methods: 372 HF patient-CP pairs will be recruited from the VA Louis Stokes (Cleveland) Healthcare System. Patients will receive automated telephone assessment and behavior change calls weekly for 12 months. For patients in both study arms, a care manager will monitor patients' assessment results via a secure website and will receive reports concerning urgent health problems by fax and pager. In the HITCM+CP group, patients' CPs also will receive tailored e-mail reports based on patients' weekly assessments. HITCM+CP patients and their CPs will use a structured protocol to review the patient's assessment results, identify self-care goals and barriers, and ensure that the patient's in-home caregivers and healthcare team remain involved. All patients and CPs will complete quantitative surveys at baseline, 6, and 12 months. The study will include a mixed-methods approach including qualitative interviews with patients, CPs and clinicians to evaluate intervention use and the service's potential for translation. The primary outcome will be HF-related quality of life at 12 months. Secondary outcomes will include self-care behavior, patient-CP relationship indicators, hospitalization, and death.

Impact: This study will evaluate a model for leveraging ICGs and structuring their role in HF patients' overall disease management. If effective, the service may provide the frequent monitoring and behavior change assistance that patients need, allowing VA to extend its impact beyond what current care management programs can realistically deliver.

ELIGIBILITY:
Inclusion Criteria:

Veterans with heart failure (HF) treated at the VA Louis Stokes (Cleveland) facilities will be eligible if they have New York Heart Association (NYHA) Class II-III diastolic or systolic HF noted by inpatient or outpatient ICD-9 codes.

Exclusion Criteria:

Veterans treated at the VA Louis Stokes (Cleveland) facilities will be ineligible if they:

* have a serious mental illness or cognitive dysfunction, e.g., psychosis, dementia, or active substance abuse (alcohol and/or other drugs);
* do not speak English fluently;
* are receiving palliative care due to advanced HF or other health problems;
* receive the majority of their HF care from providers outside of the VA;
* are unable to use a telephone to respond to weekly automated self-management support calls; or
* are unable to nominate an eligible informal caregiver.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2009-06; Primary Completion 2013-01 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. Piette, PhD, Principal Investigator — VA Ann Arbor Healthcare System
Locations (2):
- United States (2):
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - VA Medical Center, Cleveland, Cleveland, Ohio

REFERENCES:
- [Result] Piette JD, Rosland AM, Marinec NS, Striplin D, Bernstein SJ, Silveira MJ. Engagement with automated patient monitoring and self-management support calls: experience with a thousand chronically ill patients. Med Care. 2013 Mar;51(3):216-23. doi: 10.1097/MLR.0b013e318277ebf8. PMID 23222527
- [Derived] Piette JD, Striplin D, Marinec N, Chen J, Aikens JE. A randomized trial of mobile health support for heart failure patients and their informal caregivers: impacts on caregiver-reported outcomes. Med Care. 2015 Aug;53(8):692-9. doi: 10.1097/MLR.0000000000000378. PMID 26125415
- [Derived] Piette JD, Striplin D, Marinec N, Chen J, Trivedi RB, Aron DC, Fisher L, Aikens JE. A Mobile Health Intervention Supporting Heart Failure Patients and Their Informal Caregivers: A Randomized Comparative Effectiveness Trial. J Med Internet Res. 2015 Jun 10;17(6):e142. doi: 10.2196/jmir.4550. PMID 26063161

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard mHealth: Weekly IVR calls for 12 months
- mHealth Plus CarePartner: Wkly IVR calls for 12 months+feedback to CarePartner
Period: Overall Study
Arm/Group | Standard mHealth | mHealth Plus CarePartner
Started | 183 | 189
Completed | 156 | 153
Not Completed | 27 | 36

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard mHealth | mHealth Plus CarePartner | Total
Number analyzed (Participants) | 156 | 153 | 309
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 74 | 144
  >=65 years | 86 | 79 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (10.6) | 67.8 (10.6) | 68.1 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 154 | 153 | 307
Region of Enrollment [Number; unit: participants]
  United States | 156 | 153 | 309
Heart Failure-specific Quality of Life [Mean (Standard Deviation); unit: units on a scale] — Measured by the Minnesota Living with heart Failure Questionnaire (MLHFQ). Lower scores indicate better functioning. MLHFQ contains 21 items with answer choices ranging from 0 to 5. Overall scores on the instrument range from 0 to 105.
  units on a scale | 40.4 (25.1) | 41.2 (23.7) | 40.8 (24.4)
Revised Heart Failure Self-Care Behavior Scale (HFSCB) [Mean (Standard Deviation); unit: units on a scale] — Higher scores indicate better Heart Failure self-care. The HFSCB contains 29 items with answer choices ranging from 0 to 5. The total score ranges from 0 to 145.
  units on a scale | 82.9 (19.3) | 83.1 (16.3) | 83.0 (17.8)
Adherent to Heart Failure Medication [Number; unit: participants] — Number of patients with perfect Heart Failure medication adherence over the prior month as measured by the four Heart Failure Self-Care Behavior items focused on adherence.
  participants | 81 | 84 | 165

OUTCOME MEASURES:

1. Primary Outcome: Heart Failure-specific Quality of Life
Description: Measured by the Minnesota Living with Heart Failure Questionnaire (MLHFQ). Lower scores indicate better functioning. MLHFQ contains 21 items with answer choices ranging from 0 to 5. Overall scores on the instrument range from 0 to 105.
Time Frame: twelve-month followup
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- mHealth+Carepartner: Weekly IVR calls for 12 months+CarePartner feedback
Arm/Group | Standard mHealth | mHealth+Carepartner
Number analyzed (Participants) | 156 | 153
units on a scale | 37.0 (25.7) | 38.6 (24.8)
Statistical Analysis 1: Comparison: Standard mHealth vs mHealth+Carepartner; Test type: Superiority or Other; p = .975, Regression, Logistic; Mean Difference (Final Values) = .74, 95% CI 2-sided [-4.62 to 4.77], Standard Deviation 2

2. Secondary Outcome: Revised Heart Failure Self-Care Behavior Scale (HFSCB)
Description: Higher scores indicate better Heart Failure self-care. The HFSCB contains 29 items with answer choices ranging from 0 to 5. The total score ranges from 0 to145.
Time Frame: twelve-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- mHealth+Carepartner: Weekly IVR calls for 12 months+feedback to CarePartner
Arm/Group | Standard mHealth | mHealth+Carepartner
Number analyzed (Participants) | 156 | 153
units on a scale | 92.1 (18.7) | 90.5 (17.0)
Statistical Analysis 1: Comparison: Standard mHealth vs mHealth+Carepartner; Test type: Superiority or Other; p = .349, Regression, Logistic; Mean Difference (Final Values) = -1.87, 95% CI 2-sided [-5.78 to 2.05], Standard Deviation 1.7

3. Secondary Outcome: Adherent to Heart Failure Medication
Description: Percent of patients with perfect Heart Failure medication adherence over the prior month as measured by the four Heart Failure Self-Care Behavior items focused on adherence.
Time Frame: twelve-month follow-up
Measure: Number; unit: percentage of participants/perfect adher
Arm/Group | Standard mHealth | mHealth+Carepartner
Number analyzed (Participants) | 156 | 153
percentage of participants/perfect adher | 52.6 | 66.7
Statistical Analysis 1: Comparison: Standard mHealth vs mHealth+Carepartner; Test type: Superiority or Other; p = .007, Regression, Logistic; Difference in Percent = 14, 95% CI 2-sided [3.9 to 24.2], Standard Deviation 6

ADVERSE EVENTS:
Arm/Group | Standard mHealth | mHealth+Carepartner
Serious Adverse Events (participants affected / at risk) | 0/183 | 0/189
Other Adverse Events (participants affected / at risk) | 0/183 | 0/189

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes